CLINICAL TRIAL: NCT01670981
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy, Safety and Tolerability of Transendocardial Injection of Ixmyelocel-T in Subjects With Heart Failure Due to Ischemic Dilated Cardiomyopathy (IDCM).
Brief Title: An Efficacy, Safety and Tolerability Study of Ixmyelocel-T Administered Via Transendocardial Catheter-based Injections to Subjects With Heart Failure Due to Ischemic Dilated Cardiomyopathy (IDCM)
Acronym: ixCELLDCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vericel Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABI 55-1202-1
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Ischemic Dilated Cardiomyopathy (IDCM)
Keywords: Ischemic dilated cardiomyopathy; Heart failure; ixCELL; ixCELL DCM; IDCM; DCM; stem cells; MSC; cell therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ixmyelocel-T (Experimental): Ixmyelocel-T delivered by catheter-based intramyocardial injection procedure.
  Interventions: Biological: ixmyelocel-T
- Placebo (Placebo Comparator): Placebo delivered by catheter-based intramyocardial injection procedure.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ixmyelocel-T — 12-20 transendocardial injections of 0.4 mL of ixmyelocel-T per injection into the left ventricle.
  Arms: ixmyelocel-T
Other: Placebo — 12-20 transendocardial injections of 0.4 mL of vehicle control per injection into the left ventricle.
  Arms: Placebo

SUMMARY:
This study is designed to assess the efficacy, safety and tolerability of ixmyelocel-T compared to placebo (vehicle control) when administered via transendocardial catheter-based injections to patients with end stage heart failure due to IDCM, who have no reasonable revascularization options (either surgical or percutaneous interventional) likely to provide clinical benefit.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of ixmyelocel-T compared to placebo (vehicle control) on the average per patient number of all-cause deaths, cardiovascular hospital admissions, and unplanned outpatient or emergency department visits to treat acute decompensated heart failure, over the 12 months following administration of investigational product (IP).

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females;
2. Age 30 to 86 years of age;
3. Diagnosis of ischemic dilated cardiomyopathy;
4. LVEF ≤ 35% by echocardiogram;
5. Symptomatic heart failure in NYHA functional class III or IV;
6. Subject is not a candidate for reasonable revascularization procedures that will produce clinical improvement;
7. Subject is receiving appropriate clinical standard of care heart failure therapy, as tolerated and as dictated by a subject's current medical condition, for at least 30 days prior to screening;
8. Must have an automatic implantable cardioverter defibrillator (AICD);
9. Worsening heart failure hospitalization or equivalent within 6 months prior to screening, hospitalization equivalent defined as an unplanned outpatient/emergency department visit for treatment of acute decompensated heart failure; or have an N-terminal prohormone B-type natriuretic peptide (NT-proBNP) ≥2000 pg/mL or BNP ≥400 pg/mL within 30 days of screening (including screening); or have a 6-minute walk test (6MWT) distance of ≤400 meters at screening;
10. Life expectancy of at least 12 months in the opinion of the Investigator;
11. LV wall thickness ≥ 7mm (by echocardiogram) at anticipated target injection area;
12. Hemodynamic stability without IV vasopressors or support devices;
13. Given medical history and concurrent medication, subject is an acceptable candidate for bone marrow aspiration and cardiac catheterization and transendocardial injection procedures in the opinion of the Investigator;
14. Willing and able to comply scheduled visits and tolerate study procedures.
15. Voluntarily provide a personally-signed and dated informed consent.

Exclusion Criteria:

Disease-specific:

1. Severe primary valvular heart disease including, but not limited to, aortic valve stenosis and insufficiency;
2. VAD implantation, heart transplantation, cardiomyoplasty, left ventricular reduction surgery, or cardiac shunt implantation;
3. Planned heart failure-related device interventions (e.g., VAD implantation, initial cardiac resynchronization therapy) or planned cardiac procedures (e.g., heart transplant, cardiomyoplasty, valvular repair);
4. Current arrhythmias that would prohibit accurate NOGA® electromechanical mapping and NOGA®-guided injections;
5. LV thrombus (as documented on echocardiography or LV angiography);
6. Myocardial infarction, stroke or transient ischemic attack within 3 months prior to screening;
7. Percutaneous coronary intervention, valvuloplasty, cardiac surgery, and other major cardiac procedure within 30 days prior to screening;
8. In the opinion of the Investigator, the subject's left ventricular wall is unsuitable for transendocardial injections (due to thickness or other reasons).

   Medical History:
9. Stroke or transient ischemic attack (TIA) within 3 months of screening;
10. Hemoglobin A1c (HbA1c) ≥ 9% at screening;
11. Diabetic subjects with uncontrolled or untreated proliferative retinopathy as determined by dilated eye exam administered by a qualified eye care professional as per American Diabetes Association guidelines;
12. Blood clotting disorder not caused by medication (e.g., thrombophilia);
13. Active malignancy (non-basal cell) requiring surgery, chemotherapy, and/or radiation in the past 12 months;
14. Drug or alcohol abuse that would interfere with the subject's compliance with study procedures;
15. Allergies to any equine, porcine, or bovine products;
16. Body mass index (BMI) ≥ 40 kg/m2 at screening;
17. Established chronic kidney disease (CKD) requiring dialysis (Stage 5); estimated creatinine clearance < 15 mL/min at screening;
18. Subject has allergy or is unable to tolerate cardiac imaging contrast agents; also the inability to get a good quality echocardiogram image at screening (as determined by the imaging core lab).

    Laboratory Parameters:
19. Abnormal laboratory values (performed at central lab) at screening:

    * Platelets < 50,000 μL;
    * Hemoglobin < 9.0 g/dL;
    * Aspartate aminotransferase/alanine aminotransferase (AST/ALT) > 3 times the upper limit of normal (ULN);
    * Human immunodeficiency virus 1 (HIV 1), HIV 2, or syphilis positive (rapid plasma reagin [RPR]);
    * Active hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies;
    * NOTE: Additional lab tests may be performed per local requirements including but not limited to: hepatitis B core antibody, human T lymphotropic virus I/II.

    Exclusionary Procedures, Devices, or Medication:
20. Subjects receiving anti-angiogenic drugs (e.g., anti-vascular endothelial growth factor [VEGF]);
21. Chronic exposure to cytotoxic therapy for oncologic or chronic non-oncologic reasons in the prior 3 months or expected requirement over the course of the study;
22. Concurrent participation in another interventional clinical trial or receiving experimental intervention within 30 days of screening or having previously been exposed to Aastrom's ixmyelocel T product or previously received allogeneic cell therapy, autologous cell therapy cultured with animal proteins.
23. In the opinion of the Investigator, the subject is unsuitable for cellular therapy or has a food/drug allergy, surgical or medical condition, clinically significant psychiatric disorders, poor nutritional status, or lab abnormality requiring further medical evaluation that may interfere with the investigational product, interfere with the study results' interpretation, interfere with the subject's ability to complete the study or compromise the subject's safety.

Ages: 30 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Average number of clinical events over 12 months post-treatment. | 12 Months
  The primary endpoint will assess the efficacy of ixmyelocel-T compared to placebo (vehicle control) on the average number of events per patient over 12 months post-treatment in each treatment arm (total number events in each arm/total number of patients in each arm). The events include: all-cause deaths, cardiovascular hospitalizations, and unplanned outpatient or emergency department visits to treat acute decompensated heart failure. The clinical events used in this endpoint will be adjudicated by an independent clinical endpoint committee who are blinded to treatment.

SECONDARY OUTCOMES:
The win ratio of the hierarchical occurrence of all-cause deaths/left ventricular assist device (LVAD) implant/heart transplant, cardiovascular hospitalizations, and unplanned outpatient and ED interventions to treat ADHF | 12 Months
  This is a composite end point. This endpoint will be primarily assessed excluding events considered to be related to administration of IP. An analysis including IP administration-related events will also be conducted as part of the sensitivity analyses.
Change from baseline to 12 months post-treatment in 6-minute walk test. | 12 Months
  A secondary objective will be to evaluate the changes from baseline to 12 months post-treatment in the distance walked as measured by the 6-minute walk test.
Change from baseline to 12 months post-treatment in left ventricular function as evaluated by echocardiography. | 12 Months
  A secondary objective will be to evaluate the change in left ventricular function as measured by echocardiography for left ventricular ejection fraction (LVEF).
Change from baseline to 12 months post-treatment in quality of life. | 12 Months
  A secondary objective will be to evaluate the change in quality of life (total score) in patients treated with ixmyelocel-T compared to placebo using the Minnesota Living with Heart Failure Questionnaire.
Change from baseline to 12 months post-treatment in NYHA Classification. | 12 Months
  A secondary objective will be to evaluate the change from baseline to Month 12 in NYHA Classification in patients treated with ixmyelocel-T compared to placebo.
Percent of patients with adverse events. | 12 Months
  A secondary objective will be to evaluate the overall safety and tolerability of ixmyelocel-T versus placebo in patients with DCM from time of aspiration through 12 months post-treatment/follow-up by % of patients with adverse events.
Percent of patients with major adverse cardiac events (MACE). | 12 Months
  A secondary objective will be to evaluate the overall safety and tolerability of ixmyelocel-T versus placebo in patients with DCM by the percentage of patients who experience MACE events. MACE events include: unstable angina requiring hospitalization, myocardial infarction, stroke, worsening heart failure requiring hospitalization, VAD implantation, heart transplant, resuscitated sudden death, and cardiovascular death.

CONTACTS AND LOCATIONS:
Locations (36):
- United States (34):
  - Cardiology, P.C. & Center for Therapeutic Angiogenesis, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Scripps Clinic, La Jolla, California
  - UCSD Medical Center, La Jolla, California
  - Cedars-Sinai Heart and Lung Institute, Los Angeles, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - St. John's Regional Medical Center, Oxnard, California
  - Stanford University, Stanford, California
  - Cardiology Research Associates, Daytona Beach, Florida
  - University of Florida - Division of Cardiology, Gainesville, Florida
  - Mayo Clinic Florida (Jacksonville), Jacksonville, Florida
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Division of Cardiology, Boston, Massachusetts
  - Michigan CardioVascular Institute, Saginaw, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Newark Beth Israel Hospital, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - The Carl and Edyth Linder Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - University Hospitals - Case Medical Center, Cleveland, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - UPMC Cardiovascular Institute, Pittsburgh, Pennsylvania
  - Veterans Administration Healthcare System, Pittsburgh, Pennsylvania
  - Stern Cardiovascular Foundation, Inc., Germantown, Tennessee
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - Methodist DeBakey Heart and Vascular Center, Houston, Texas
  - University of Utah Health Services Center, Salt Lake City, Utah
  - Swedish Medical Center - Cherry Hill Professional Building, Seattle, Washington
  - University of Wisconsin-Madison Cardiovascular Medicine, Madison, Wisconsin
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Montreal Heart Institute, Montreal, Quebec

REFERENCES:
- [Derived] Patel AN, Henry TD, Quyyumi AA, Schaer GL, Anderson RD, Toma C, East C, Remmers AE, Goodrich J, Desai AS, Recker D, DeMaria A; ixCELL-DCM Investigators. Ixmyelocel-T for patients with ischaemic heart failure: a prospective randomised double-blind trial. Lancet. 2016 Jun 11;387(10036):2412-21. doi: 10.1016/S0140-6736(16)30137-4. Epub 2016 Apr 5. PMID 27059887
- See also: Vericel Corporation Homepage — http://www.vcel.com/